CLINICAL TRIAL: NCT04453540
Title: Impact of the Syndromic PCR System FilmArray on Management of ICU Patients With Severe Pulmonary Disease in the Context of the Covid-19 Pandemic.
Brief Title: FilmArray and Management of ICU Patients With Pneumonia in the Covid-19 Context
Acronym: FAP-REA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Reims University hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI101
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Infectious Disease; Pneumonia; Molecular Diagnosis; Covid-19; Antibiotic Stewardship
MeSH Terms: conditions — Communicable Diseases; Pneumonia; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FilmArray PCR on respiratory samples — Molecular test performed on respiratory samples realized for microbiological routine testing as part of the care

SUMMARY:
The research aims to determine the impact of a syndromic mutiplex PCR assay (FilmArray) on the management of patients hospitalized in ICU for severe respiratory disease.

During the SARS-CoV-2 outbreak, the diagnosis of pneumonia has become considerably more complex as the biological, radiological and clinical criteria of covid-19 interfere with the standard criteria for the diagnosis of severe respiratory diseases. Moreover, patients with COVID-19 are at higher risk of developing other associated infections and thus, patients have therefore often been treated with antibiotics, adequately or not, due to difficulty to quickly identify the etiology of their symptoms with conventional methods.

In order to improve their treatment, both diagnostic and therapeutic, we set up a new syndromic molecular test in our laboratories to accelerate and improve the pneumonia management and antibiotic stewardship. This research will include 100 to 150 adult patients hospitalized in ICU during the first half of 2020. It will take place within the Nancy University Hospital and the Reims University Hospital, France.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years affiliated to a social security system
* Patients who have received complete information about the research and who have not objected to the use of its data
* Patients with suspected SARS-Cov-2 infection
* Patients for which a FilmArray test has been realized on its respiratory samples between 1st of March and 1st of July 2020.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in ICU at the hospitals of Nancy and Reims for severe respiratory diseases during the first half of 2020
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic decision | 24 h following the FilmArray results
  Antibiotic prescription modification following the FilmArray results as:
  * No prescription
  * No change in antibiotic utilization
  * Antibiotic initiation
  * Antibiotic escalation
  * Antibiotic de-escalation
  * Antibiotic discontinuation

REFERENCES:
- [Derived] Novy E, Goury A, Thivilier C, Guillard T, Alauzet C. Algorithm for rational use of Film Array Pneumonia Panel in bacterial coinfections of critically ill ventilated COVID-19 patients. Diagn Microbiol Infect Dis. 2021 Nov;101(3):115507. doi: 10.1016/j.diagmicrobio.2021.115507. Epub 2021 Jul 23. PMID 34364096